# Clinical Trial of Solriamfetol for Excessive Sleepiness Related to Shift Work Disorder

ClinicalTrials.gov ID: NCT04788953

Document Date: January 13, 2025

Subject Identification

General Consent Form Template Version Date: January 2019

Protocol Title: Clinical Trial of Solriamfetol for Excessive Sleepiness related

to Shift Work Disorder

Principal Investigator: Charles A. Czeisler, Ph.D., M.D.

Site Principal Investigator:

Description of Subject Population: Early Morning Workers, age 18-64

### About this consent form

Please read this form carefully. It tells you important information about a research study. A member of our research team will also talk to you about taking part in this research study. People who agree to take part in research studies are called "subjects." This term will be used throughout this consent form.

Partners HealthCare System is made up of Partners hospitals, health care providers, and researchers. In the rest of this consent form, we refer to the Partners system simply as "Partners."

If you decide to take part in this research study, you must sign this form to show that you want to take part. We will give you a signed copy of this form to keep.

# **Key Information**

Taking part in this research study is up to you. You can decide not to take part. If you decide to take part now, you can change your mind and drop out later. Your decision won't change the medical care you get within Partners now or in the future.

The following key information is to help you decide whether or not to take part in this research study. We have included more details about the research in the Detailed Information section that follows the key information.

# Why is this research study being done?

In this research study we want to learn more about whether the medication solriamfetol improves daytime sleepiness in workers who start work at very early times (between 3 and 7am).

How long will you take part in this research study?


IRB Protocol No: 2021P000509 IRB Expiration Date: 1/13/2026
Consent Form Valid Date: 1/13/2025 IRB Submission: CR4/AME30




If you decide to join this research study, it will take you about 8 weeks to complete the study. During this time, we will ask you to make a total of 6 study visits. Four of those visits will be to the Ambulatory Clinical Center (ACC) at 221 Longwood Avenue. Two of the visits will be to the Center for Clinical Investigation (CCI) at Brigham and Women's Hospital at 75 Francis Street. Those two visits will last approximately 8-10 hours each.

### What will happen if you take part in this research study?

If you decide to join this research study, the following things will happen. You will undergo a screening process, including an all-night home sleep test, to see if you are healthy enough to take part in the study. If we find you meet the study criteria, you will be scheduled for a baseline study visit to test your daytime sleepiness. That lasts for 8-10 hours, and consists of a series of four nap tests. If you meet the study criteria on this baseline visit, you can then begin the study. For 2 weeks you will wear an activity monitor on your wrist all the time (24/7) and fill out a daily diary about your work and sleep habits. At the end of the 2 weeks you will come for a study visit where you will receive 2 weeks of study medication. For the next 2 weeks you will continue to wear the activity monitor and keep a daily diary, and in addition you will take the study medication each morning before you go to work. After 2 weeks you will come for another study visit and receive 2 more weeks of study medication. For the next 2 weeks you will continue to wear the activity monitor and keep a daily diary, and take the study medication each morning before you go to work. After a total of 4 weeks taking the study medication you will come for a second nap study visit About a week after the second nap study, we will ask you to come back for final brief visit where we can give you a physical exam and check to see how you are doing.

# Why might you choose to take part in this study?

We cannot promise any benefits to you from taking part in this research study. However, possible benefits may include improvement in your daytime sleepiness, which may thereby improve your overall functioning. Others with Shift Work Disorder may benefit in the future from what we learn in this study.

# Why might you choose NOT to take part in this study?

Taking part in this research study has some risks and requirements that you should consider carefully.

People taking monoamine oxidase (MAO) inhibitors should not take part in this study. Important risks and possible discomforts from the study medication include headache, nausea, decreased appetite, anxiety, and insomnia.

IRB Expiration Date: 1/13/2026 IRB Submission: CR4/AME30




A detailed description of side effects, risks, and possible discomforts can be found later in this consent form in the section called "What are the risks and possible discomforts from being in this research study?".

Other things to consider are the number and frequency of study visits.

## What other treatments or procedures are available for your condition?

Other treatments or procedures that are available to treat Shift Work Disorder include changing work hours, taking naps to increase sleep time, or using caffeine or prescription wake-promoting drugs such as modafinil (Provigil®) or armodafinil (Nuvigil®).

# If you have questions or concerns about this research study, whom can you call?

You can call us with your questions or concerns. Our telephone numbers are listed below. Ask questions as often as you want.

Charles A. Czeisler, PhD, MD is the person in charge of this research study. You can call him at 617-732-4013 M-F 9-5. You can also call Jeanne Duffy, MBA, PhD at 617-732-7995 M-F 10-6 or Kirsi-Marja Zitting, PhD at 617-525-8339 M-F 10-6 with questions about this research study.

If you have questions about the scheduling of appointments or study visits, call the Study Coordinator at 617-525-8657.

If you want to speak with someone **not** directly involved in this research study, please contact the Partners Human Research Committee office. You can call them at 857-282-1900.

You can talk to them about:

- Your rights as a research subject
- Your concerns about the research
- A complaint about the research
- Any pressure to take part in, or to continue in the research study

Subject Identification


## **Detailed Information**

A description of this clinical trial will be available on *http://www.ClinicalTrials.gov*, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### Why is this research study being done?

We are doing this research study to find out if solriamfetol (Sunosi®) can help people with Shift Work Disorder (excessive daytime sleepiness due to the timing of work hours) feel more alert when they work early morning shifts.

Solriamfetol (Sunosi®) is approved by the U.S. Food and Drug Administration (FDA) to treat excessive daytime sleepiness in Obstructive Sleep Apnea and Narcolepsy, but solriamfetol (Sunosi®) is not approved by the FDA to treat Shift Work Disorder.

This research study will compare solriamfetol to placebo. The placebo looks exactly like solriamfetol, but contains no solriamfetol. During this study you may get a placebo instead of solriamfetol. Placebos are used in research studies to see if the results are due to the study drug or due to other reasons.

# Who will take part in this research?

We are asking you to take part in this research study because you describe having the symptoms of Shift Work Disorder. Shift Work Disorder occurs in individuals who work nontraditional hours like split shifts, graveyard shifts, early morning shifts, or rotating shifts. It is characterized by excessive sleepiness, lack of refreshing sleep, and drowsiness. These symptoms can affect both work time and free time.

About 500 people will be enrolled in this study at Brigham and Women's Hospital (BWH) in order to find 100 subjects who can complete the study.

Axsome Therapeutics, Inc. is paying for this research to be done.

# What will happen in this research study?

If you choose to take part in this study, we will ask you to sign this consent form before we do any study procedures.

### **Screening Visit (Visit 1)**

The Screening Visit will take place at 221 Longwood Avenue and will take about 3 hours. At this visit, we will review and sign this consent form and then do some tests and procedures to see




if you qualify to take part in this research study. The study doctor will review the results of these tests and procedures, but some results will not be available until a few days after the visit. If you don't qualify, the study doctor will tell you why. We may do the consent form review and signing by phone or video call. We may ask you to fill out some of the screening questionnaires online using a computer.

At this visit, we will:

- Ask you about your medical history
- Do a physical exam, including height, weight, blood pressure, and heart rate
- Draw 3 blood samples
- Ask you for a urine sample
- Test your urine for certain drugs
- Test your urine for pregnancy, if you are a female able to become pregnant. Pregnant women cannot take part in this research study.
- Do an ECG (electrocardiogram)
- Ask you to fill out some questionnaires about your general health and well-being, sleep habits, work schedule, mental and emotional health, and mood
- Have you take home a Home Sleep Test device to use that night or the next night while you are sleeping

### **Urine Drug Screen**

During this study, we will test your urine for certain drugs such as cannabis/marijuana, including illegal drugs, e.g., cocaine, opiates, phencyclidine (PCP), amphetamines. We will also test your urine for alcohol. If your urine shows you have taken any of these substances or drugs, you can't be in this study. The results of the urine drug test will not become part of your medical record. These test results will, however, remain part of your study record.

#### ECG (electrocardiogram)

This test checks the electrical activity of your heart. We will place several small, sticky pads on your chest, arms, and legs. Each pad has a wire attached. The wires connect to a machine that makes a recording of your heart rhythm. This painless test takes about 15 minutes.

### **Home Sleep Test**

After we have received the results from the tests done in the Screening Visit, we will have you take a Home Sleep Test. The test lasts all night while you are sleeping and is to see if you have any sleep problems that you do not know about.

• You will wear a sleep monitor one night. The monitor records information about your breathing, how well your body is getting oxygen, your leg movements, and how often you wake up. You will put it on just before going to bed, and take it off as soon as you get up. You will be given instructions on how to use it.




- The monitor has two soft elastic belts that you will wear while you sleep. You will place one around your chest and the other around your waist to measure your breathing. You will also put a sensor near your nose to measure your breathing. You will put a sensor on your finger to measure the oxygen level in your blood. You will also place one or two sensors on your lower legs to measure if your legs move while you sleep. You may also be asked to place a sensor on your forehead and another behind your ear to measure the number of times you wake up. All these sensors will stay on you during the whole night while you sleep.
- You will also be asked to complete a brief questionnaire to record the timing, duration, and quality of your sleep on the night you wore the sleep equipment.
- You will be asked to return the sleep monitor and the questionnaire to study staff, either in person or via FedEx or another courier company. We will give you a box to send the sleep monitor back to us.
- You may be asked to re-do the Home Sleep Test if we do not get a good recording.

### Baseline Visit (Visit 2) – Nap Study

Visit 2 will take place in the main hospital building at 75 Francis Street and will take about 10 hours. At this visit, we will:

- Ask you to arrive at or shortly before the time you usually begin work
- Take your vital signs (temperature, heart rate, blood pressure)
- Ask you to fill out some questionnaires about your work productivity, sleepiness, and ability to get things done, as well as your mood and other symptoms
- Have you meet with study personnel to answer questions about your work hours and sleepiness
- Have you take part in a series of four 40-minute naps (about every two hours) to test how sleepy you are
- Ask you to self-rate your sleepiness right before each nap

### Nap Test

When you arrive for Visit 2 we will place a series of sensors on your face and scalp so we can record your EEG (brain waves), eye movements, and muscle activity, and two sensors on your chest to measure your EKG. To take these measurements, a staff member will clean your skin with alcohol and then put small electrodes (sensors) on the skin of your scalp and face. There will be 4 to 8 sensors on your head and 5 to 7 on your face. We will put the sensors on your head with a special glue. We will put the sensors on your face with tape. We will put two sensors on your chest to measure your heart rate. All these sensors will remain on you for the entire visit.

As soon as the sensors are all on, you will take the first of four naps. For each nap we will:

- Ask you to use the bathroom
- Pull down blackout shades in your room (if your room has windows)





- Ask you to turn off any devices you have with you and to give us your mobile phone to keep outside your room
- Ask you to get into bed
- Ask you to rate your sleepiness on a 9-point scale
- Turn out all the lights in your room except a small nightlight
- Ask you to try to remain awake as long as you can

If you fall asleep, we will come into the room to wake you up, the nap will be ended, and you will be asked to get out of bed until the next scheduled nap. If you do not fall asleep after 40 minutes, we will end the nap opportunity and you will be asked to get out of bed until the next scheduled nap.

There will be a total of four naps, each about two hours apart. In between the naps you will be offered a breakfast and a lunch, you will be asked to fill out some questionnaires and meet with study staff, but you will otherwise have some free time to read, watch a movie, or do other sedentary activities in your study room.

After the fourth nap is over, we will remove all the sensors and the visit will be over. If you meet the study criteria, you can begin the Baseline Segment of the study.

## **Baseline Segment**

The Baseline Segment lasts 2 weeks and is carried out at home. During this time we will:

- Give you an activity monitor to wear on your wrist the entire 2 weeks, 24/7.
- Ask you to fill out a sleep and work diary every day during the 2 weeks.

### **Randomization Visit (Visit 3)**

Visit 3 will be scheduled at the end of the 2-week Baseline Segment and will take place at 221 Longwood Avenue. It will take about 1 hour. At this visit, we will:

- Take your temperature, blood pressure, and heart rate
- Test your urine for pregnancy, if you are a female able to become pregnant. Pregnant women cannot take part in this research study.
- Review the activity data from your activity monitor and the entries in your sleep and work diary with you
- Ask you to tell us about any symptoms you have had and ask you questions about how your mental and emotional health and mood have been

If you still qualify for the study, we will assign you by chance (like a coin toss) to the solriamfetol group or the placebo group. You and the study doctor cannot choose your study group. You will have an equal chance of being assigned to the solriamfetol group.




You and the study doctor won't know which study group you are in, but he can find out if necessary.

### **Randomization Segment 1**

This part of the study will last 2 weeks and is carried out at home. During this time we will:

- Have you continue to wear an activity monitor on your wrist the entire 2 weeks, 24/7.
- Have you continue to fill out a sleep and work diary every day during the 2 weeks.
- Take the study drug.
- Have a short phone or video appointment at the end of the first week of this segment.

### **Taking the Study Drug**

We will give you a 2-week supply of the study drug to take home with you.

### **Your Study Diary**

The sleep and work diary will have additional questions about the study drug. You will write down the time you take the study drug, how much study drug you take, and whether you have any side effects.

After one week, we will schedule a brief phone or video appointment with you. This appointment will take about half an hour. During this appointment we will:

• Ask you to tell us about any symptoms you have had and ask you questions about how your mental and emotional health and mood have been

#### Visit 4

Visit 4 will be scheduled at the end of the 2-week Randomization Segment 1 and will take place at 221 Longwood Avenue. It is like Visit 3, and will take about 1 hour. At this visit, we will:

- Take your temperature, blood pressure, and heart rate
- Review the activity data from your activity monitor and the entries in your sleep and work diary with you
- Ask you to tell us about any symptoms you have had and ask you questions about how your mental and emotional health and mood have been
- Give you another 2-week supply of the study drug

### **Randomization Segment 2**

This part of the study will last 2 weeks and is carried out at home. It is the same as Randomization Segment 1. During this time we will:

- Have you continue to wear an activity monitor on your wrist the entire 2 weeks, 24/7.
- Have you continue to fill out a sleep and work diary every day during the 2 weeks.
- Take the study drug by mouth when you first wake up on the mornings when you have an early morning work shift.





• Have a short phone or video appointment at the end of the first week of this segment.

### Visit 5 – Nap Study

Visit 5 is scheduled at the end of the 2 weeks of Randomization Segment 2. Visit 5 will take place in the main hospital building at 75 Francis Street and will be like Baseline Visit 2, lasting about 10 hours. At this visit, we will carry out all the same procedures as in Visit 2. In between the naps, we will also carry out some of the procedures from the Screening visit, including:

- Do a physical exam, including height, weight, blood pressure, and heart rate
- Draw 2 blood samples
- Ask you for a urine sample
- Do an ECG (electrocardiogram)
- Ask you to fill out some of the same questionnaires about your general health and wellbeing, sleep habits, work schedule, mental and emotional health, and mood that you filled out during screening
- Ask you to tell us about any symptoms you have had and ask you questions about how your mental and emotional health and mood have been

After the fourth nap is over, we will remove all the sensors, take back the activity monitor, and the visit will be over. We will schedule a follow-up visit for about one week later.

### Follow-up Phase (Visit 6)

About one week after you stop taking the study drug and complete the second Nap Visit, you will come in for one follow-up visit (Visit 6). This visit will take place at 221 Longwood Avenue. It is like Visits 3 and 4, and will take about 1 hour. At this visit, we will:

- Do a physical exam, including height, weight, blood pressure, and heart rate
- Ask you to tell us about any symptoms you have had and ask you questions about how your mental and emotional health and mood have been

### **After You Complete the Study**

After you complete the study, we will refer you back to your own doctor for your ongoing medical care.

### **Stopping the Study Early**

If you decide to stop taking part in the study for any reason, we will ask you to make a final study visit. You will need to return all unused study drug, the activity monitor, and your study diary at this visit. If you have completed 1 or more weeks of taking the study drug, we will ask you to do a Nap visit for this final visit, which will take about 10 hours. At this visit, we will carry out all the activities normally done in Visit 5.




If you stop taking part in the study at an earlier point, the final study visit will take about 1 hour. At this visit, we will:

- Do a physical exam, including height, weight, blood pressure, and heart rate
- Draw 2 blood samples
- Ask you for a urine sample
- Do an ECG (electrocardiogram)
- Ask you to fill out some of the same questionnaires about your general health and wellbeing, sleep habits, work schedule, mental and emotional health, and mood that you filled out during screening
- Ask you to tell us about any symptoms you have had and ask you questions about how your mental and emotional health and mood have been

Also, the study doctor may take you out of the study without your permission. This may happen because:

- The study doctor thinks it is best for you to stop taking the study drug
- You can't make the required study visits
- The Funding Agency decides to stop the study
- We stop doing the study for other reasons

If this happens, the study doctor will explain why you need to stop taking part in the study. We will ask you to come in for a final study visit as described above.

# Review of Medical Records from Hospital Admissions or Emergency Department Visits

Partners has an electronic system that lets your study doctors know if you are admitted to a Partners Hospital, or if you visit a Partners Hospital Emergency Department. We want to make sure the study doctors know about any possible problems or side effects you experience while you are taking part in the study.

### Study Information Included in Your Electronic Medical Record

A notation that you are taking part in this research study may be made in your electronic medical record. Information from the research that relates to your general medical care may be included in the record (for example: list of allergies, results of standard blood tests done at the hospital labs).

Please ask your study doctor if you have any questions about what information will be included in your electronic medical record.

# How may we use and share your samples and health information for other research?





The information we collect in this study may help advance other research. If you join this study, we may remove all information that identifies you (for example, your name, medical record number, and date of birth) and use these de-identified samples and data in other research. It won't be possible to link the information or samples back to you. Information and/or samples may be shared with investigators at our hospitals, at other academic institutions or at for-profit, commercial entities. You will not be asked to provide additional informed consent for these uses.

# Will you get the results of this research study?

You and your doctor should not expect to get information about the results of the research study or the results of your individual participation in the research study. We will study samples and information from many people. It could take many years before anyone knows whether the results have any meaning. There is a small chance that we could find out something from the study that might be important to your health. If this happens, we may contact you to find out if you would like to learn more. However, even if we find something important to your health, we cannot guarantee that you will be contacted.

# What are the risks and possible discomforts from being in this research study?

### **Risks of Taking Solriamfetol**

Taking solriamfetol may cause you to have one or more of the side effects listed below.

Common side effects:

- Headache (10 out of 100 people reported this side effect)
- Nausea (4 out of 100 people reported this side effect)
- Decreased appetite (4 out of 100 people reported this side effect)
- Anxiety (3 out of 100 people reported this side effect)
- Insomnia (3 out of 100 people reported this side effect)

Less common side effects (fewer than 2 out of 100 people reported these side effects):

- Rapid heart beat
- Dry mouth
- Constipation
- Irritability
- Increased blood pressure
- Increased heart rate
- Diarrhea

Uncommon side effects:

Subject Identification


- Agitation, restlessness
- Bruxism
- Cough
- Chest discomfort, pain
- Excessive sweating
- Restlessness
- Thirst
- Weight loss

There may be other risks of solriamfetol that are currently unknown.

As with any drug, an allergic reaction can occur. Allergic reactions can be mild or more serious, and can even result in death. Common symptoms of an allergic reaction are rash, itching, skin problems, swelling of the face and throat, or trouble breathing. If you think you are having an allergic reaction, call the study doctor right away. If you are having trouble breathing, call 911 immediately.

### Risks to an Embryo or Fetus, or to a Breastfeeding Infant

The effect of solriamfetol on an embryo or fetus (developing baby still in the womb), or on a breastfeeding infant, is unknown and may be harmful. Because of these unknown risks, women cannot take part in this study if they are:

- Pregnant
- Trying to become pregnant
- Breastfeeding

If you are a menopausal woman and have not had a menstrual period for the past 12 months or more, you will not need to have a pregnancy test. Also, if you have had any well-documented method of surgical sterilization, you will not need to have a pregnancy test. Methods of surgical sterilization include having had a hysterectomy (removal of the uterus), bilateral oophorectomy (removal of both ovaries), a tubal ligation (having your tubes tied), and transvaginal occlusion (plugging the opening of the tubes with a coil). All other female subjects must have a negative pregnancy test before starting the study drug.

If you are sexually active and able to become pregnant, you must agree to use one of the birth control methods listed below. You must use birth control **for the entire study and for at least** 30 days after your last dose of study drug.

Acceptable birth control methods for use in this study are:

 hormonal methods, such as birth control pills, patches, injections, vaginal rings, or implants




- intrauterine device (IUD)
- abstinence (no sex)

If you miss a period, or think you might be pregnant during the study, you must tell the study doctor immediately. If you become pregnant, you must stop taking the study drug and stop taking part in the study. The study doctor may ask you to join a registry of patients who have become pregnant while taking this study drug.

If you are sexually active and able to father a child, you must agree to use one of the birth control methods listed below. You must use birth control for the entire study and for at least 30 days after your last dose of study drug. You must also agree to not donate sperm for the entire study and for at least 30 days after your last dose of study drug.

Acceptable birth control methods that you can use in this study are:

- condoms
- abstinence (no sex)

Acceptable birth control methods that your partner(s) should use are:

- hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants
- intrauterine device (IUD)

#### **Risks of Blood Draws**

You may have a bruise (a black and blue mark) or pain where we take the blood samples. There is also a small risk of infection, lightheadedness, and/or fainting. The total amount of blood drawn in the study will be less than 30 mL. This is about 6 teaspoons of blood. There should be no risks to your health from giving this much blood.

### **Text Messages**

Text messages by mobile/cell phones are a common form of communication. If you previously indicated that you would like to receive text messages that are relevant to the research study, we may send you text messages during the study, and we want to inform you of the potential risks. Texting over mobile/cell phones carries security risks because text messages to mobile/cell phones are not encrypted. This means that information you send or receive by text message could be intercepted or viewed by an unintended recipient, or by your mobile/cell phone provider or carrier.

Below are some important points about texting in this research study.




- •Text messages are not encrypted, and therefore carry security risks. This research study and Mass General Brigham are not responsible for any interception of messages sent through unencrypted text message communications.
- •You will be responsible for all fees charged by your carrier's service plan for text messaging. This research study and Mass General Brigham are not responsible for any increased charges, data usage against plan limits or changes to data fees from the research texts (Include language if participants are paid/given stipends to cover potential charges).
- •Text messages will only be read during regular business hours. Texts sent on nights or weekends will not be read until the next business day.
- •Text messaging should not be used in case of an emergency. If you experience a medical emergency, call 911 or go to the nearest hospital emergency department.
- •You may decide to not send or receive text messages with staff associated with this research study at any time. You can do this in person or by sending the research number a text message that says "Stop Research Text."
- •Your agreement applies to this research study only. Agreeing to other texts from Mass General Brigham, for example appointment reminders, is a separate process. Opting out of other texts from Mass General Brigham is a separate process as well.
- •It is your responsibility to update your mobile/cell phone number with this research study in the event of a change.

# What are the possible benefits from being in this research study?

You may not benefit from taking part in this research study. If you receive solriamfetol, it is possible that your excessive daytime sleepiness due to early morning shifts will improve while you are taking it. However, because solriamfetol is not FDA-approved for this disorder, your doctor cannot prescribe it after you finish the study.

Others with excessive daytime sleepiness due to early morning shifts may benefit in the future from what we learn in this study.

# What other treatments or procedures are available for your condition?

You do not have to take part in this study to be treated for excessive daytime sleepiness or Shift Work Disorder. Other treatments or procedures that are available to treat the excessive sleepiness from Shift Work Disorder include:

- modafinil (brand name Provigil)
- armodafinil (brand name Nuvigil)
- caffeine or other stimulants



General Template Version Date: December 2008

# Can you still get medical care within Partners if you don't take part in this research study, or if you stop taking part?

Yes. Your decision won't change the medical care you get within Partners now or in the future. There will be no penalty, and you won't lose any benefits you receive now or have a right to receive.

We will tell you if we learn new information that could make you change your mind about taking part in this research study.

# What should you do if you want to stop taking part in the study?

If you take part in this research study, and want to drop out, you should tell us. We will make sure that you stop the study safely. We will also talk to you about follow-up care, if needed.

Also, it is possible that we will have to ask you to drop out of the study before you finish it. If this happens, we will tell you why. We will also help arrange other care for you, if needed.

# Will you be paid to take part in this research study?

You will be paid \$150.00 for completing all the screening procedures, including the phone prescreen, the Informed Consent visit, the screening questionnaires, the Screening Visit (Visit 1), and the Home Sleep Test.

You will receive \$ 420.00 per week for wearing the wrist activity monitor 24/7, completing the daily sleep-work-drug diary, and coming for the study visits. This includes the 2 weeks of the Baseline Segment (and Visit 3), the 2 weeks of Randomization Segment 1 (and Visit 4), and the 2 weeks of Randomization Segment 2 (total \$2,520).

You will receive \$ 350.00 for completing each of the Nap Studies (Visits 2 and 5; total \$700 .00).

For completing all study visits, returning all study equipment and materials, and completing the Follow-up Visit (Visit 6), you will receive \$2,630.





If you complete the entire study you will receive a total of \$6,000. If you do not complete the entire study you will be compensated for what you have completed, but you will not receive any Follow-up Visit "end of study" payment.

We will give you a voucher or reimburse you up to \$15.00 for parking at 221 Longwood Avenue for Visits 1, 3, 4 and 6.

For Visits 2 and 5 (the Nap Studies) we will pay for the cost of your transportation up to \$50 (\$25/each way).

We may use your samples and information to develop a new product or medical test to be sold. The Sponsor, hospital, and researchers may benefit if this happens. There are no plans to pay you if your samples or information are used for this purpose.

# What will you have to pay for if you take part in this research study? Axsome Therapeutics is providing the study drug at no cost.

Study funds will pay for certain study-related items and services. We may bill your health insurer for, among other things, routine items and services you would have received even if you did not take part in the research. You will be responsible for payment of any deductibles and copayments required by your insurer for this routine care or other billed care. If you have any questions about costs to you that may result from taking part in the research, please speak with the study doctors and study staff. If necessary, we will arrange for you to speak with someone in Patient Financial Services about these costs.

# What happens if you are injured as a result of taking part in this research study?

We will offer you the care needed to treat any injury that directly results from taking part in this research study. We reserve the right to bill your insurance company or other third parties, if appropriate, for the care you get for the injury. We will try to have these costs paid for, but you may be responsible for some of them. For example, if the care is billed to your insurer, you will be responsible for payment of any deductibles and co-payments required by your insurer.

Injuries sometimes happen in research even when no one is at fault. There are no plans to pay you or give you other compensation for an injury, should one occur. However, you are not giving up any of your legal rights by signing this form.





If you think you have been injured or have experienced a medical problem as a result of taking part in this research study, tell the person in charge of this study as soon as possible. The researcher's name and phone number are listed in the beginning of this consent form.

# If you take part in this research study, how will we protect your privacy?

Federal law requires Partners to protect the privacy of health information and related information that identifies you. We refer to this information as "identifiable information."

### In this study, we may collect identifiable information about you from:

- Past, present, and future medical records
- Research procedures, including research office visits, tests, interviews, and questionnaires

# Who may see, use, and share your identifiable information and why they may need to do so:

- Partners researchers and staff involved in this study
- The sponsor(s) of the study, and people or groups it hires to help perform this research or to audit the research
- Other researchers and medical centers that are part of this study
- The Partners ethics board or an ethics board outside Partners that oversees the research
- A group that oversees the data (study information) and safety of this study
- Non-research staff within Partners who need identifiable information to do their jobs, such as for treatment, payment (billing), or hospital operations (such as assessing the quality of care or research)
- People or groups that we hire to do certain work for us, such as data storage companies, accreditors, insurers, and lawyers
- Federal agencies (such as the U.S. Department of Health and Human Services (DHHS) and agencies within DHHS like the Food and Drug Administration, the National Institutes of Health, and the Office for Human Research Protections), state agencies, and foreign government bodies that oversee, evaluate, and audit research, which may include inspection of your records
- Public health and safety authorities, if we learn information that could mean harm to you or others (such as to make required reports about communicable diseases or about child or elder abuse)


IRB Protocol No: 2021P000509 IRB Expiration Date: 1/13/2026
Consent Form Valid Date: 1/13/2025 IRB Submission: CR4/AME30




#### • Other:

Some people or groups who get your identifiable information might not have to follow the same privacy rules that we follow and might use or share your identifiable information without your permission in ways that are not described in this form. For example, we understand that the sponsor of this study may use your identifiable information to perform additional research on various products or conditions, to obtain regulatory approval of its products, to propose new products, and to oversee and improve its products' performance. We share your identifiable information only when we must, and we ask anyone who receives it from us to take measures to protect your privacy. The sponsor has agreed that it will not contact you without your permission and will not use or share your identifiable information for any mailing or marketing list. However, once your identifiable information is shared outside Partners, we cannot control all the ways that others use or share it and cannot promise that it will remain private.

Because research is an ongoing process, we cannot give you an exact date when we will either destroy or stop using or sharing your identifiable information. Your permission to use and share your identifiable information does not expire.

The results of this research study may be published in a medical book or journal, or used to teach others. However, your name or other identifiable information **will not** be used for these purposes without your specific permission.

## **Your Privacy Rights**

You have the right **not** to sign this form that allows us to use and share your identifiable information for research; however, if you don't sign it, you can't take part in this research study.

You have the right to withdraw your permission for us to use or share your identifiable information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing. Once permission is withdrawn, you cannot continue to take part in the study.

If you withdraw your permission, we will not be able to take back information that has already been used or shared with others, and such information may continue to be used for certain purposes, such as to comply with the law or maintain the reliability of the study.

You have the right to see and get a copy of your identifiable information that is used or shared for treatment or for payment. To ask for this information, please contact the person in charge of this research study. You may only get such information after the research is finished.


IRB Protocol No: 2021P000509 IRB Expiration Date: 1/13/2026
Consent Form Valid Date: 1/13/2025 IRB Submission: CR4/AME30

General Consent Form Template

Version Date: January 2019

Subject Identification

# **Informed Consent and Authorization**

# **Statement of Person Giving Informed Consent and Authorization**

- I have read this consent form.
- This research study has been explained to me, including risks and possible benefits (if any), other possible treatments or procedures, and other important things about the study.
- I have had the opportunity to ask questions.
- I understand the information given to me.

# Signature of Subject:

| I give my consent to take part in this research study and agree to allow my health information be used and shared as described above. | | |
|---|---|---|
| Subject | Date | Time (optional) |
| Signature of Study Doctor or Person C | Obtaining Cons | ent: |
| Statement of Study Doctor or Person Obtain | ing Consent | |
| <ul> <li>I have explained the research to the stud</li> <li>I have answered all questions about this</li> </ul> | • | the best of my ability. |
| Study Doctor or Person Obtaining Consent | Date | Time (optional) |
| Consent Form Version: 16 October 2023 | | |

